CLINICAL TRIAL: NCT00895050
Title: Impact of the Use of a Computer-based Tools on the Clinical Management and Evolution of Patients With Rheumatoid Arthritis.
Brief Title: Study Evaluating Impact of the Use of a Computer-based Tool on the Clinical Management of RA Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Other Study IDs: 0881X1-4576; B1801084
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed with RA
  Interventions: Other: Review of clinical records

INTERVENTIONS:
Other: Review of clinical records

SUMMARY:
The primary purpose of this study is to evaluate a computer-based tool on the clinical management of patients with rheumatoid arthritis in Spain.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria:

* Patients, male or female, over 18 years old.
* Patients diagnosed with RA according to investigator criteria
* Patients with a disease evolution >= 1 year
* Patients with > = 5 affected joints

Exclusion Criteria:

Exclusion Criteria:

* Patients with other muscle skeletal, rheumatic and/or degenerative diseases different from RA.
* Patients who are taking part or have taken part in a clinical trial or in a study with drugs within the last 12 months. Any condition that, in the investigator's judgment would interfere with the subject's ability to comply with protocol requirements or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA treated in rheumatology offices
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Global mean DAS28 at 6 and at 12 months of follow-up. Differences between global mean DAS28 at 6 and at 12 months compared to baseline | 12 months

SECONDARY OUTCOMES:
Disease activity (DAS28; number affected joints; CRP; ESR; PGA).-Number of variables used in patient's follow-up; number of treatment adjustments. -Investigator's satisfaction with the computer-based tool (specific questionnaire) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4576&StudyName=Study%20Evaluating%20%20Impact%20of%20the%20Use%20of%20a%20Computer-based%20Tool%20on%20the%20Clinical%20Management%20of%20RA%20Patients